CLINICAL TRIAL: NCT04109794
Title: Comparison of Two Techniques in Gingival Recession Treatment. One-year Clinical Follow-up Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, H. Gencay Keceli, Associate Professor, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SerdarEvginer
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-CTG (Active Comparator): Envelope connective tissue graft
  Interventions: Procedure: E-CTG
- SCAF (Active Comparator): Semilunar connective tissue graft
  Interventions: Procedure: E-CTG

INTERVENTIONS:
Procedure: E-CTG — Envelope connective tissue graft

SUMMARY:
42 patients were treated either with E-CTG (N=20) or SCAF (N=22). The recordings included clinician-based (recession depth, recession width, probing depth, clinical attachment level, keratinized tissue width, tissue thickness, clinical attachment gain (CAG), root coverage (RC), keratinized tissue change (KTC)) and patient-based (wound healing index (WHI), dentine hypersensitivity (DH), tissue appearance, patient expectations and aesthetics) parameters that were taken at baseline, T1 (sixth week), T2 (sixth month) and T3 (first year).

ELIGIBILITY:
Inclusion Criteria:

* single Miller I GR defects ≤3mm at upper anterior or premolar teeth
* systemically healthy
* identifiable cemento-enamel junction (CEJ)
* PD ≤3 mm

Exclusion Criteria:

* periodontal surgery experience in the past two years
* excessive contacts
* mobility
* caries
* loss of vitality
* smoking
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
recession depth | baseline
  Distance between CEJ and GM
recession depth | 6 weeks
  Distance between CEJ and GM
recession depth | 6 months
  Distance between CEJ and GM
recession depth | 12 months
  Distance between CEJ and GM

SECONDARY OUTCOMES:
recession width | baseline
  horizontal distance between two borders of recession at CEJ level
recession width | 6 weeks
  horizontal distance between two borders of recession at CEJ level
recession width | 6 months
  horizontal distance between two borders of recession at CEJ level
recession width | 12 months
  horizontal distance between two borders of recession at CEJ level
probing depth | baseline
  distance between GM and base of gingival sulcus
probing depth | 6 weeks
  distance between GM and base of gingival sulcus
probing depth | 6 months
  distance between GM and base of gingival sulcus
probing depth | 12 months
  distance between GM and base of gingival sulcus
clinical attachment level | baseline
  distance between CEJ and base of gingival sulcus
clinical attachment level | 6 weeks
  distance between CEJ and base of gingival sulcus
clinical attachment level | 6 months
  distance between CEJ and base of gingival sulcus
clinical attachment level | 12 months
  distance between CEJ and base of gingival sulcus
keratinized tissue width | baseline
  distance between GM and MGJ
keratinized tissue width | 6 weeks
  distance between GM and MGJ
keratinized tissue width | 6 months
  distance between GM and MGJ
keratinized tissue width | 12 months
  distance between GM and MGJ

REFERENCES:
- [Derived] Evginer MS, Olgun E, Parlak HM, Dolgun AB, Keceli HG. Comparison of two techniques in gingival recession treatment: A randomized one-year clinical follow-up study. Dent Med Probl. 2022 Jan-Mar;59(1):121-130. doi: 10.17219/dmp/137621. PMID 35394710